CLINICAL TRIAL: NCT03414112
Title: Investigating the Impact of Oxytocin on the Neurobiological Underpinnings of Socioemotional Deficits in Anorexia Nervosa
Brief Title: The Impact of Oxytocin on the Neurobiology of Anorexia Nervosa
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Klarman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PSYCH-2017-26002
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Participants with anorexia nervosa and age-matched control participants will complete two separate fMRI and test meal assessments: one following administration of intranasal oxytocin and one following placebo. The study will be double blind.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double blind; participants and study staff will not know if the participant is receiving intranasal oxytocin or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Oxytocin Placebo (Placebo Comparator): Intranasal placebo
  Interventions: Biological: Intranasal oxytocin
- Intranasal Oxytocin (Experimental): Intranasal oxytocin
  Interventions: Biological: Intranasal oxytocin

INTERVENTIONS:
Biological: Intranasal oxytocin — oxytocin is a peptide hormone that influences social affiliation

SUMMARY:
This study will use a randomized, controlled, double-blind design involving the administration of intranasal oxytocin (INOT) or placebo to adults with anorexia nervosa, restricting subtype and age-matched controls prior to neuroimaging to assess the impact on frontolimbic brain activity in response to socioemotional stimuli as well as eating behavior in a test meal paradigm.

DETAILED DESCRIPTION:
The primary objective of this investigation is to determine the impact of oxytocin (OT), a peptide hormone that influences social affiliation, on socioemotional neural circuitry and eating disorder behavior in anorexia nervosa (AN). Because socioemotional processing deficits appear to play a key role in AN, OT is implicated as a potential biological mechanism by which eating disorder behavior (e.g., restrictive eating) is maintained. Used as a probe, intranasal oxytocin (INOT) provides an innovative method for examining the short-term impact of OT on socioemotional neural processing disturbances and eating disorder behavior in AN. The proposed study tests a theoretical model of the role of OT in the maintenance of AN by using an INOT probe to determine, and potentially alter, neurobiological responses to socioemotional stimuli. Specifically, this study will use a randomized, controlled, double-blind design involving the administration of INOT or placebo to adults with AN restricting subtype and age-matched controls prior to neuroimaging to assess the impact on frontolimbic brain activity in response to socioemotional stimuli. The potential impact of INOT on restrictive eating will also be assessed in a subsequent test meal. We predict that for participants with AN, INOT, but not placebo, will normalize frontolimbic activation in response to social reward stimuli and prefrontal activation in response to social threat stimuli. In addition, the investigators predict that AN participants will display reduced restrictive eating in a test meal paradigm following INOT (but not placebo) administration. Finally, investigators predict that changes in restrictive eating following INOT administration will be mediated by altered frontolimbic responding to socioemotional cues. This investigation will provide an essential link uniting the data supporting the importance of socioemotional processing deficits in AN with the emerging role of INOT in altering the neural circuits involved in social behavior to test an innovative neurobiological maintenance model of AN.

ELIGIBILITY:
Inclusion Criteria:

* All participants:

  1. Age > 18 years old
  2. Female (given the potential sex differences to endogenous OT to INOT)
  3. Ability to read and speak in English
  4. Right-handed
* Anorexia nervosa participants:

  1. DSM-5 diagnosis of AN, restricting subtype (established by the SCID-5-RV),
  2. BMI < 18.5 kg/m2 within the past month

     Exclusion Criteria:

     All participants

  <!-- -->

  1. Medical instability or current pregnancy or lactation
  2. Current substance use disorder, psychosis, or bipolar-I disorder
  3. Contraindication for fMRI (e.g., implanted metal)
  4. History of neurological disorder/injury (e.g., stroke; head injury with > 10 minutes loss of consciousness)
  5. Food allergy that cannot be accommodated through substitutions to the laboratory test meal
  6. Lacking capacity to consent
  7. Contraindications for intranasal oxytocin administration
  8. Acute suicidality
  9. Psychoactive medication (e.g., antidepressants, antipsychotics)

     Exclusion for participants without anorexia nervosa

  <!-- -->

  1. Current DSM-5 Axis-I diagnosis or current or past eating disorder diagnosis
  2. BMI < 19.0

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Test meal | Following intranasal oxytocin or placebo (within 1-3 hours)
  Participants will complete a test meal
fMRI measures | Following intranasal oxytocin or placebo administration (within 1-3 hours)
  Neural activation in regions of interest (ROIs) in socioemotional circuitry (i.e., ACC, amygdala, medial PFC, NAcc) in response to INOT or placebo and social threat vs. neutral tasks and social reward vs. neutral stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Carol B Peterson, PhD, Principal Investigator — University of Minnesota; Ann F Haynos, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - Dept of Psychiatry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided